CLINICAL TRIAL: NCT03622918
Title: Comparison of Efficacy and Safety of Colistin-rifampin Combination and Colistin Monotherapy in Extensively Drug-resistant Acinetobacter Baumannii: Utility of the Synergy Test Results (E-test) in Vitro
Brief Title: Colistin-rifampin Combination and Colistin Monotherapy in Extensively Drug-resistant Acinetobacter Baumannii
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Min Kwang Byun, Assisstant Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3-2016-0125
Record Dates: First submitted 2018-07-30; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Colistin; Rifampin; Acinetobacter Infections
MeSH Terms: conditions — Acinetobacter Infections | interventions — Colistin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- colistin monotherapy (Sham Comparator): The subjects will be treated with colistin monotherapy. Colistin (100 mg, colistin sodium methanesulfonate, SCD Pharm., Seoul, Korea) will be intravenously administered with 100 mL of normal saline with 8 hours interval. Treatment should be maintained daily administration for at least 7 days and up to 28 days. Duration of antibiotics treatment will be determined through discussion by pulmonology and infection specialist.
  Interventions: Drug: colistin monotherapy
- colistin-rifampin combination (Experimental): The subjects will be treated with colistin and rifampin combination therapy. Colistin (100 mg, colistin sodium methanesulfonate, SCD Pharm., Seoul, Korea) will be intravenously administered with 100 mL of normal saline with 8 hours interval. Rifampin (600 mg, rifampin, Yuhan, Seoul, Korea) will be orally administered daily. Treatment should be maintained daily administration for at least 7 days and up to 28 days. Duration of antibiotics treatment will be determined through discussion by pulmonology and infection specialist.
  Interventions: Drug: colistin and rifampin combination therapy

INTERVENTIONS:
Drug: colistin and rifampin combination therapy — Colistin (100 mg, colistin sodium methanesulfonate, SCD Pharm., Seoul, Korea) will be intravenously administered with 100 mL of normal saline with 8 hours interval. Rifampin (600 mg, rifampin, Yuhan, Seoul, Korea) will be orally administered daily. Treatment should be maintained daily administration for at least 7 days and up to 28 days. Duration of antibiotics treatment will be determined through discussion by pulmonology and infection specialist.
  Other Names: colistin/rifampin combination therapy
  Arms: colistin-rifampin combination
Drug: colistin monotherapy — . Colistin (100 mg, colistin sodium methanesulfonate, SCD Pharm., Seoul, Korea) will be intravenously administered with 100 mL of normal saline with 8 hours interval. Treatment should be maintained daily administration for at least 7 days and up to 28 days. Duration of antibiotics treatment wil be determined through discussion by pulmonology and infection specialist .
  Arms: colistin monotherapy

SUMMARY:
The investigators aimed to confirm the utility of the synergy test results (E-tesT) in vitro to predict the efficacy and safety of colistin-rifampin combination and colistin monotherapy in extensively drug-resistant acinetobacter baumannii.

DETAILED DESCRIPTION:
We will searched pneumonia patients with CoRAB in Gangnam Severance Hospital. Subjects will be enrolled and randomized in a blinded fashion using a computerized random number generator (permuted-block randomization) for treatment with colistin and rifampin combination and colistin only at a ratio of 1:1. We will perform the E-test MIC:MIC ratio method to predict in vitro synergy of colistin and rifampin combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pneumonia, blood septicemia, urinary tract infection, or other infection or even colonization with evidence of extensively drug-resistant Acinetobacter baumannii infection

Exclusion Criteria:

* Hypersensitivity reaction to colistin or rifampin
* use of colistin or rifampin in 15 days prior to screening
* evidence of extensively drug-resistant Acinetobacter baumannii infection in 15 days prior to screening
* CLcr < 15 mL/min, ALT or AST > 3xULN, total bilirubin > 2xULN, Hb < 7 gm/dL, ANC < 500/mm3, Platelet < 50,000/mm3

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2017-09-24 (Actual); Study Completion 2018-06-21 (Actual)

PRIMARY OUTCOMES:
microbiologic response | 14 days
  negative conversion of culture study (eradication)

SECONDARY OUTCOMES:
clinical response | 14 days
  clinical resolution of fever, symptoms and infectious sign
mortality | 30 days
  mortality

IPD SHARING:
Plan to Share IPD: Undecided
in discuss

REFERENCES:
- [Derived] Park HJ, Cho JH, Kim HJ, Han SH, Jeong SH, Byun MK. Colistin monotherapy versus colistin/rifampicin combination therapy in pneumonia caused by colistin-resistant Acinetobacter baumannii: A randomised controlled trial. J Glob Antimicrob Resist. 2019 Jun;17:66-71. doi: 10.1016/j.jgar.2018.11.016. Epub 2018 Nov 23. PMID 30476654